CLINICAL TRIAL: NCT03958630
Title: PET Imaging of Neuroinflammation in Neurodegenerative Diseases Via a Novel TSPO Radioligand
Brief Title: PET Imaging of Neuroinflammation in Neurodegenerative Diseases Via a Novel Translocator Protein (TSPO) Radioligand
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI closed the protocol due to low recruitment
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 190095; 19-M-0095
Record Dates: First submitted 2019-05-21; First posted 2019-05-22 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-01

CONDITIONS: Dementia
Keywords: Fronto Temporal Dementia; Amyloid; Neuroinflammation
MeSH Terms: conditions — Dementia; Alzheimer Disease; Neuroinflammatory Diseases | interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole; Positron-Emission Tomography; Radionuclide Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Healthy volunteers (Experimental): Participants underwent brain positron emission tomography (PET) scan with [11C]ER176 and/or [11C]PIB followed by brain magnetic resonance imaging (MRI)
  Interventions: Drug: 11C-ER176; Drug: 11C-PIB; Diagnostic Test: Positron Emission Tomography (PET) Scan
- Subjects with chromosome 9 open reading frame 72 (C9ORF72) (Experimental): Participants underwent brain positron emission tomography (PET) scan with [11C]ER176 and/or [11C]PIB followed by brain magnetic resonance imaging (MRI)
  Interventions: Drug: 11C-ER176; Drug: 11C-PIB; Diagnostic Test: Positron Emission Tomography (PET) Scan
- Subjects with Frontotemporal dementia (FTD) (Experimental): Participants underwent brain positron emission tomography (PET) scan with [11C]ER176 and/or [11C]PiB followed by brain magnetic resonance imaging (MRI)
  Interventions: Drug: 11C-ER176; Drug: 11C-PIB; Diagnostic Test: Positron Emission Tomography (PET) Scan

INTERVENTIONS:
Drug: 11C-ER176 — PET biomarker for inflammation
Drug: 11C-PIB — PET biomarker for amyloid
Diagnostic Test: Positron Emission Tomography (PET) Scan — Participants underwent PET scan with [11C]ER176 and/or 11C-PIB

SUMMARY:
Background:

Aging-related progressive neurological disorders include frontotemporal dementia, Lou Gehrig s disease, and Alzheimer s disease. Little is known about what causes these disorders. Brain inflammation may be involved. Researchers want to see if scans using radioactive drugs can show brain inflammation.

Objective:

To see if the drug [11C]ER176 can show inflammation in the brain in people with certain progressive neurological disorders compared to healthy adults. Also to find genes that might be associated with or cause these disorders.

Eligibility:

People ages 18 and older with an aging-related neurological disorder, and healthy adults

Design:

Participants will be screened with a medical history, physical exam, neurological exam, psychiatric history, and blood tests.

Participants will have 2-5 visits for the first session. They will have 2 PET scans and 1 MRI scan. They may have 3 more sessions: 6 months to about 18 months later, 1 year after that, and about 30 months to 5 years after the first visit. There may be up to 20 total visits.

For the scans, participants will lie on a bed that slides into the scanners. For the PET scans, a strap will fix their head in place. A radioactive drug will be injected through a catheter. A needle will guide a thin plastic tube into an arm vein. Additional catheters may be put in place to draw blood. Each PET will take 2 hours. The MRI will take 30 60 minutes.

At each session, participants will have a brief interview, medical history, physical exam, blood and urine tests, heart tests, and memory and thinking tests. They may donate blood for DNA tests.

DETAILED DESCRIPTION:
Objectives

The primary objective is to explore if human subjects with neurodegenerative diseases exhibit different level of neuroinflammation, as measured by brain uptake of a 3rd generation [11C]ER176 TSPO ligand, compared to control subjects. The secondary objectives are to determine, 1) if [11C]ER176 TSPO brain uptake shows disease-specific patterns across different neurodegenerative diseases and/or genetic mutations, and 2) if longitudinal imaging of individual patients shows a correlation between interval change of tracer uptake and disease progression.

Study population

Adults referred with a clinical diagnosis or with an increased risk of frontotemporal dementia, amyotrophic lateral sclerosis, Alzheimer s disease, other related adult-onset neurodegenerative disorders, or healthy control subjects.

Design

Participants will undergo a general and neurological exam, a standard battery of neuropsychological tests to measure cognitive function, blood tests for analysis of TSPO polymorphisms, MRI of the brain, and PET imaging with the [11C]ER176 TSPO radioligand and [11C]PIB amyloid radioligand. Participants will be invited to return for repeat evaluations approximately 1, 2, and 3-5 years after their initial evaluation.

Outcome measures

Brain PET and MRI scans will be co-registered for anatomic definition of regions of interest, and standard uptake value (SUV) will be calculated in various brain regions. [11C]ER176 PET data will be analyzed with compartmental modeling. [11C]PIB PET and MRI data will be adjunctly used for segregating the collected data by disease subtype. For the primary objective, we will compare TSPO radioligand uptake of healthy controls compared to subjects with neurodegenerative diseases. For secondary objectives, we will determine if neuroanatomical regions of tracer uptake differ across different neurodegenerative disease subtypes, and if interval change of tracer uptake correlates with disease progression in longitudinal imaging of individual subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients will be included if they
* Are age 18 or older

  * Have the ability to understand and sign an informed consent, or have a DPA or a court-appointed guardian (or be able to understand the DPA process to appoint a DPA) to provide consent for adults without consent capacity
  * Have been given a diagnosis by a neurologist of frontotemporal dementia, frontotemporal lobar degeneration, primary progressive aphasia, semantic dementia, motor neuron disorder, amyotrophic lateral sclerosis, primary lateral sclerosis, progressive bulbar palsy, corticobasal syndrome, Huntington disease, Alzheimer s disease, or other related adult-onset neurodegenerative disease

    2. Subjects with an increased risk of neurodegenerative diseases will be included if they
  * Are age 18 or older
  * Are able to give written informed consent
  * Have known family history or other risk of an adult-onset genetic neurodegenerative disease, and/or mutation in a gene known to cause an adult-onset neurodegenerative disease

    3. Healthy subjects will be included if they
  * Are age 18 or older
  * Are willing and able to complete all study procedures
  * Are able to give written informed consent
  * Are medically healthy
  * Are enrolled in 01-M-0254 The Evaluation of Participants with Mood and Anxiety Disorders and Healthy Volunteers (PI: Dr. Carlos Zarate) or 17-M-0181, Recruitment and Characterization of Healthy Research Volunteers for National Institute of Mental Health (NIMH) Intramural Studies (PI: Dr. Joyce Chung)

EXCLUSION CRITERIA:

1. Patients or subjects with an increased risk of neurodegenerative diseases will be excluded if they

   * Have other major neurological or medical diseases that may cause progressive weakness or cognitive dysfunction, such as structural brain or spinal cord disease, metabolic diseases, paraneoplastic syndromes, infectious diseases, peripheral neuropathy or radiculopathy or other significant neurological abnormalities
   * Have an unstable medical condition that, in the opinion of the investigators, makes participation unsafe (e.g., active infection or untreated malignancy)
   * Require daytime ventilator support at the time of study entry
   * Are unable to travel to NIH
   * Have recent exposure to radiation related to research (e.g., PET from other research) that, when combined with this study, would be above the allowable limits
   * Have inability to lie flat and/or lie still on camera bed for at least two hours, including claustrophobia, overweight greater than the maximum for the scanner, and uncontrollable behavioral symptoms, which will be screened by an interview with patient and/or caregiver during the screening visit
   * Are pregnant or breastfeeding
   * Participants must not have substance use disorder or alcohol use disorder. However, alcohol or cannabis use by themselves are not exclusion criteria, unless that use impairs function
   * Are unable to have an MRI scan (e.g., pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pumps, or shrapnel fragments, metal fragments in the eye)
   * NIMH employees/staffs or NIH employees who are subordinates/relatives/co-workers of investigators
2. Healthy subjects will be excluded if they

   * Have any history of medical illness or injury with the potential to affect study data interpretation or to be any medical contraindication to the procedures performed in the study, including active infection and untreated malignancy.
   * Have clinically significant laboratory abnormalities based on test performed under screening protocol 01-M-0254 or 17-M-0181
   * Have recent exposure to radiation related to research (e.g., PET from other research) that, when combined with this study, would be above the allowable limits
   * Have inability to lie flat on camera bed for at least two hours, including claustrophobia and overweight greater than the maximum for the scanner
   * Are pregnant or breastfeeding
   * Participants must not have substance use disorder or alcohol use disorder. However, alcohol or cannabis use by themselves are not exclusion criteria, unless that use impairs function
   * Are unable to have an MRI scan (e.g., pacemakers or other implanted electrical devices, brain stimulators, dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pumps, or shrapnel fragments, metal fragments in the eye)
   * NIMH employees/staffs or NIH employees who are subordinates/relatives/co-workers of investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2023-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Innis, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-M-0095.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Volunteers | Subjects With Chromosome 9 Open Reading Frame 72 (C9ORF72) | Subjects With Frontotemporal Dementia (FTD)
Started | 6 | 3 | 4
Completed | 6 | 3 | 2
Not Completed | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Withdrawn due to the 2019 pandemic | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers | Subjects With Chromosome 9 Open Reading Frame 72 (C9ORF72) | Subjects With Frontotemporal Dementia (FTD) | Total
Number analyzed (Participants) | 6 | 3 | 4 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 3 | 9
  >=65 years | 3 | 0 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 3 | 10
  Male | 1 | 1 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 5 | 3 | 4 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 3 | 4 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Standard Uptake Value Ratio Compared to the Cerebellum (SUVR) Area Under the Curve (AUC) (60-90min)
Description: Participants underwent brain positron emission tomography (PET) scan with [11C]ER176 and standard uptake value (SUV) was measured over 90 minutes and divided by SUV of the cerebellum to determine difference of [11C]ER176 brain uptake
Time Frame: Up to 90 minutes during scan
Population: All participants who completed the PET scan
Measure: Mean (Standard Deviation); unit: SUV Ratio (SUVR)
Arm/Group | Healthy Volunteers | Subjects With Frontotemporal Dementia (FTD) | Subjects With Chromosome 9 Open Reading Frame 72 (C9ORF72)
Number analyzed (Participants) | 6 | 2 | 3
SUV Ratio (SUVR)
  Dorsolateral Prefrontal Cortex | 1.154816988 (0.1068451736460) | 1.243023793 (0.20560563) | 0.936561195 (0.190544723)
  Dorsomedial Prefrontal Cortex | 0.996700383 (0.071340712) | 0.989731836 (0.093928709) | 0.905523672 (0.048246962)
  Orbitofrontal Lobe | 1.217485758 (0.088415727) | 1.267286508 (0.045403115) | 1.047192088 (0.146706043)
  Perisylvian Cortex, Left | 1.143352336 (0.102185733) | 1.132367538 (0.049940532) | 1.029305407 (0.066022192)
  Perisylvian Cortex, Right | 1.090685411 (0.071228603) | 1.112003017 (0.09381086) | 0.941024006 (0.055892402)
  Parietal Lobe, Left | 1.073048863 (0.083878696) | 1.034142945 (0.01253728) | 0.918176888 (0.114668223)
  Parietal Lobe, Right | 1.020202657 (0.069903326) | 1.031347183 (0.03211946) | 0.848570905 (0.190475917)
  Medial Temporal Lobe, Left | 1.08451324 (0.07643309) | 1.064745227 (0.093063402) | 1.032603069 (0.036960689)
  Medial Temporal Lobe, Right | 1.080818839 (0.054571041) | 1.126409887 (0.037945068) | 1.006852539 (0.041618527)
  Lateral Temporal Lobe, Left | 1.000872064 (0.095177072) | 1.009331898 (0.006341876) | 0.928285311 (0.046290454)
  Lateral Temporal Lobe, Right | 0.970093545 (0.056699904) | 0.953890974 (0.022213838) | 0.868920257 (0.052268097)
  Temporal Pole, Left | 1.174033153 (0.144718189) | 1.105735482 (0.006722645) | 0.951727887 (0.184135923)
  Temporal Pole, Right | 1.083264223 (0.089675769) | 1.133115055 (0.117352842) | 0.869347972 (0.213594461)
  Occipital Lobe | 1.054680093 (0.054134358) | 1.029642393 (0.019495596) | 0.971346796 (0.048140098)
  Basal Ganglia + Thalamus | 1.005308052 (0.120193318) | 1.000347379 (0.046553725) | 0.991325953 (0.017050753)

ADVERSE EVENTS:
Time Frame: Up to 24 hours after each clinic visit for PET scan and MRI
Arm/Group | Healthy Volunteers | Subjects With Chromosome 9 Open Reading Frame 72 (C9ORF72) | Subjects With Frontotemporal Dementia (FTD)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/4

LIMITATIONS AND CAVEATS:
Secondary outcomes were not analyzed because:

* No data for the disease specific uptake across neurodegenerative diseases
* No longitudinal data was collected because the protocol was terminated due to low recruitment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/30/NCT03958630/Prot_SAP_000.pdf